CLINICAL TRIAL: NCT06558162
Title: The Effect of Two Different Self-Assessment Methods for Fetal Movement Monitoring on Maternal Psychosocial Status
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Neriman Guducu, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PR0478R1
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Fetal Movement; Mental Health Issue
Keywords: pregnancy; fetal movements; mindfetalness

STUDY DESIGN:
Intervention Model Description: Pregnant women included in the study were randomized into two groups. One group will have fetal movements assessed using the Sadovsky method. The other group will use the Mindfetalness method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Pregnant women assigned to groups will not know which method (name) they are using. The person who will conduct the research analyses will be someone independent of the researchers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfetalness Group (Experimental): The method is based on noting the quality of perceived movements, which develops maternal awareness of the health of the foetus. The method requires the mother to lie on her left side while her baby is awake and for 15 minutes focus on exactly how the baby moves, taking into account the strength, type and frequency of movement. However, the number of fetal movements is not counted during this time.
  It is also very important to understand the attitudes of the pregnant women, because a positive attitude may improve the perception of the pregnant woman and thus increase compliance with the method, whereas a negative attitude may hinder compliance with the method. Therefore, it will be important to create a positive attitude during the counselling of pregnant women in this group.
  Interventions: Behavioral: Mindfetalness
- Sadovsky Group (Active Comparator): This method involves counting the movements over a set period of time (usually 30 minutes to 2 hours). The mother should count the fetal movements at the same time every day. In this counting technique, mothers are especially asked to count after 3 meals during the day. Fetal movements are usually active in the evening. During the counting process, the mother should make sure that the baby is awake and should be calm, resting, eating, using the toilet, lying on her side and placing her hands on her abdomen. When the mother perceives the first movement of the baby, she should start recording on the monitoring chart given to her and continue counting and recording until the 10th movement is completed. If she counts less than 10 movements in the first 30 minutes, she should continue recording.
  Interventions: Behavioral: Sadovsky

INTERVENTIONS:
Behavioral: Mindfetalness — They will be instructed to lie on their left side and focus on the fetal movements for 15 minutes every day while the foetus is awake. They will also be instructed to monitor the character, strength and frequency of fetal movements (not to count them) and to seek medical advice if they feel any change in this pattern.
  After two weeks, the pregnant women will be invited back to the organisation for a follow-up interview to check whether they have performed the practice and recorded correctly. An interview will be conducted again after four weeks.
  Arms: Mindfetalness Group
Behavioral: Sadovsky — They will be asked to continue this procedure every morning, noon or evening for one month (depending on the movements of the pregnant woman and her baby, the time will be left to the pregnant woman, but it should be at the same time every day). Since the aim of the study is to increase maternal awareness rather than to determine fetal well-being, mothers will be asked to count at least 10 movements based on the "count to ten" and "Sadovsky" method, and will be asked to record the start and completion time of the movements each time. A follow-up will be made after two weeks and a final follow-up will be made after one month
  Arms: Sadovsky Group

SUMMARY:
Antenatal care is essential for a successful delivery, a healthy baby and a happy mother. The main aim of antenatal care is to take appropriate interventions to assess, protect and improve maternal and fetal health during pregnancy. There are many methods to assess fetal health during pregnancy, such as ultrasonography (USG) and non stress test (NST). Along with these methods, maternal perception and counting of fetal movements is the only method that can be easily used by the mother without the need for clinicians or equipment. When a pregnant woman begins to feel fetal movements, it is one of the first signs of fetal life and is considered an indicator of fetal well-being. Decrease or absence of fetal movements has been stated to be an important parameter in the assessment of fetal health and may be associated with the risk of intrauterine fetal death. Therefore, feeling and counting of fetal movements is the basis for the assessment of fetal health.

DETAILED DESCRIPTION:
Two methods are recommended for the identification of fetal movements. These are the Cardiff method and the Sadovsky method. In the assessment of fetal health, not only the number of movements per unit of time is important, but also the strength and nature of these movements. To take this into account, in 2012 Radestad introduced another method of observing the character of the movement, called "Mindfetalness". The method is based on women who develop maternal awareness of the health of the foetus and note the quality of the perceived movements. The method requires the mother to lie on her left side while her baby is awake and focus for 15 minutes on exactly how the baby is moving, taking into account the strength, type and frequency of movement. However, the number of fetal movements is not counted during this time period. This method, which helps women to note fetal movements in order to minimise and/or eliminate adverse birth outcomes, is also reported to cause unnecessary stress to the mother, as with other methods.Although there are studies reporting that counting fetal movements contributes to maternal attachment by increasing the possibility of connecting with the unborn baby, there are also studies that found no difference in maternal-fetal attachment scores. However, it is thought that focusing on the quality rather than the quantity of movements will increase the opportunity to connect with the fetus.

There is no previous comparison in the literature between a self-assessment method that focuses on qualitative variables and a counting method to measure fetal movements. Although there is one study that used both methods, this study did not differentiate between experimental and control groups, but used the crossover method and tested both methods on the same pregnant women. Therefore, our study was planned to determine the effect of fetal movement counting with two different self-assessment methods on prenatal attachment and psychosocial status.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Over 18 years of age
* Single pregnancy
* Being between 28-32 weeks of gestation
* Primiparity
* At least primary school graduation
* No diagnosed problems related to the health of the fetus (such as fetal anomaly, intrauterine growth retardation) No risky pregnancy (such as pre-eclampsia, diabetes, heart disease, placenta previa, oligohydramnios)

Exclusion Criteria:

* Not having any disabilities that may prevent communication (speech, hearing, mental)
* No chronic or psychiatric illness
* Conception with assisted reproductive techniques

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Attachment | Pretest, Follow-up after two weeks, Follow-up after four weeks
  Prenatal Maternal Attachment Scale: Each item of the scale, which has a total of 19 items, focuses on the feelings, attitudes and behaviors of the pregnant woman towards the fetus. The scale is Likert-type and each item is scored between 1-5. Before the total score is calculated, 11 items in the scale are scored in the reverse direction. The total score for the scale is obtained by adding the scores given to all items. A high score indicates a high degree of attachment.
Stress | Pretest, Follow-up after two weeks, Follow-up after four weeks
  Perceived Stress Scale-10: The ASÖ-10 is a two-factor, with each item being rated on a 5-point Likert-type scale with response options ranging from 0 (never) to 4 (very often). The responses are reversed and the scores of the four positive items are summed over the 10 items to obtain a total score. This score ranges from 0 to 40, with higher scores indicating higher perceived stress.
Anxiety | Pretest, Follow-up after two weeks, Follow-up after four weeks
  State-Trait Anxiety Inventory: It consists of a total of forty items, including a State Anxiety Scale consisting of twenty items and a Trait Anxiety Scale consisting of twenty items. There are two types of expressions in the scales: direct and reversed. The total score obtained from each scale is between a minimum of 20 and a maximum of 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Risk perception | Pretest, Follow-up after two weeks, Follow-up after four weeks
  Risk Perception in Pregnancy Scale: It consists of nine items and 2 factors. There is a 0-100 mm linear line immediately below each item on the scale, indicating "no risk" and "extremely high risk". The total score of the scale is found by adding the scores for each of the nine items and dividing the resulting score by 9. The scale has no cut-off point. As the score obtained from the scale increases, it is accepted that the perception of risk related to the pregnant woman and her baby increases.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman Güdücü, Dr., Study Director — Kırklareli University
Locations (1):
- Neriman Güdücü, Kırklareli, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No such plans have been made as the work is still in progress